CLINICAL TRIAL: NCT00486967
Title: Insulin Resistance: A New Target in Heart Failure
Brief Title: Insulin Resistance : Heart Failure
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Other Study IDs: MAT001
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Congestive Heart Failure; Heart Failure
Keywords: Insulin resistance, heart failure, congestive heart failure,; Peak VO2, Endothelial Function, Leptin, TNF.
MeSH Terms: conditions — Heart Failure; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Heart Failure: CHF patients were identified from inpatients as well as patients attending outpatient clinics and from the general practice in the community. Diagnosis of CHF was based on the European Society of Cardiology guidelines for CHF. All patients with stable CHF were included in the study. Inpatients with CHF who were hospitalized were also included, except patients with acutely decompensated CHF requiring intravenous therapy. CHF patients with a previous diagnosis of diabetes mellitus were excluded from the study.
- Controls: A group of healthy subjects were also studied. They were recruited from the community and were clinically healthy based on history, physical examination, and blood laboratory results and were not taking any medication.

SUMMARY:
Whether insulin resistance common among Chronic Heart Failure (CHF) patients in Tayside and identify factors associated with insulin resistance in CHF.

We also want to identify mechanism for the impaired exercise capacity and reduced peak VO2 in CHF

DETAILED DESCRIPTION:
There is increasing evidence of a reciprocal interrelationship between chronic heart failure (CHF) and insulin resistance (IR). Studies have shown that patients with CHF have IR and that the degree of IR is associated with reduced exercise capacity and peak oxygen consumption (VO2).

IR has also been linked to decreased exercise capacity in patients with diabetes mellitus and other chronic disease states, as well as in healthy subjects confirming that IR is independently linked to exercise intolerance studies have shown that IR is pathophysiologically linked with CHF and is implicated in the disease progression in CHF. This is likely because IR is associated with endothelial dysfunction, inflammation, increased oxidative stress and myocardial remodelling; processes that accelerate the progression of disease in CHF. Therefore, the IR has now emerged as a potential target for intervention in improving the symptoms and outcome in patients with CHF.

However, there are still some key unanswered questions. Firstly, what is the prevalence of IR in the cohort of CHF patients in Tayside? Previous studies outside the UK examining prevalence of IR in CHF were conducted in the pre-B-blocker era. However, B-blockers, which may worsen metabolic control, are now widely used in the treatment of CHF. It is likely that the prevalence might be higher in our present cohort of patients with CHF. Secondly, what are the potential contributory factors to IR in CHF?The exact mechanisms of IR in CHF are not known. Sympathetic over-activity in CHF can acutely reduce insulin sensitivity and it also decreases the release of insulin from the pancreatic beta cells, and increases hepatic glucose production. Other mediators include cytokines and adiponectin and leptin. The loss of skeletal muscle bulk and impaired endothelial function with reduced skeletal muscle blood flow may also contribute to IR in CHF. Determining the relative importance of these various factors may help identify therapeutic strategies in overcoming IR in CHF. Finally, what is the mechanism for the impaired exercise capacity and reduced peak VO2 in CHF? Exercise VO2 measures the total body's oxygen consumption which reflects both cardiac output and peripheral utilization of oxygen. We do not know whether the problem is due to a worsening of the reduced cardiac output in CHF and/or decreased peripheral utilization. To determine this, we plan to measure the cardiac output at the same as the measurement of VO2.

The aims and objectives of the study are:

Primary objectives

* To establish the prevalence of Insulin resistance (IR) among chronic heart failure (CHF) patients in Tayside
* To identify factors associated with IR in CHF

Secondary Objectives IR could have potential functional consequences

* Is it associated with a decrease in exercise capacity ?
* Is it associated with altered endothelial function ?

Investigations:

Patients will arrive in the research laboratory having fasted overnight. Following written informed consent, patients will undergo a complete medical examination and bloods (40 ml) will be drawn for measurement of neurohormones. Thereafter, the following tests will be done:

(i). Measurement of insulin resistance will be assessed using empirical fasting insulin resistance index (FIRI).For this test fasting blood glucose and insulin level will be measured. Fasting insulin resistance index is consist of the product of plasma insulin and glucose, FIRI= fasting glucose X fasting insulin / 25.

(ii). Anthropometric measurements (for measurement of fat mass and fat free mass). Body fat can be measured by (height, weight, skin fold thickness, waist, and hip circumference). Estimation of body fat in this study will be by skin fold thickness measurement or Holtain skin fold caliper18. Measurement can use from 3 to 9 different standard anatomical sites around the body. The right side is usually only measured, by pinching the skin at the appropriate site to raise a double layer of skin and the underlying adipose tissue, but not the muscle. The calipers are then applied 1 cm below and at right angles to the pinch, and a reading taken 2 seconds later. The mean of two measurements should be taken. If the two measurements differ greatly, a third should then be done, then the median value taken. In this study the Holtain skin fold calliper will be used for measuring triceps skin fold until their two exactly similar consecutive readings from each subject.

(iv). Endothelial function will be determined by reactive hyperaemia-peripheral arterial tonometry [RH-PAT] RH-PAT is a non-invasive technique to assess peripheral microvascular endothelial function by measuring changes in digital pulse volume during reactive hyperaemia 21-24. Bonetti and colleagues21 recently reported that it is reliable non-invasive tool to identify individuals with coronary microvascular endothelial dysfunction digital. The device (Itamar Medical Ltd., Caesarea, Israel) consists of two finger-mounted probes, which include a system of inflatable latex air cushions within a rigid external case. The probe design allows the application of a constant and evenly distributed near-diastolic counter pressure within the entire probe, which increases sensitivity by unloading arterial wall tension, and prevents venous blood pooling to avoid venoarteriolar reflex vasoconstriction. Pulsatile volume changes of the fingertip are sensed by a pressure transducer and transferred to a personal computer where the signal is band pass-filtered (0.3 to 30 Hz), amplified, displayed, and stored.

The PAT studies will perform with the patient in the supine position and both hands on the same level in a comfortable, thermoneutral environment. A blood pressure cuff will be placed on one upper arm (study arm), while the contralateral arm serves as a control (control arm); RH-PAT probes will be placed on one finger (finger II, III, or IV) of each hand (same finger on both hands). The fingers on either side of the one with the probe will be separated using soft sponge rings, and continuous recording of pulsatile blood volume responses from both hands will be initiated. After a 10-min equilibration period, the blood pressure cuff on the study arm will be inflated to 60 mm Hg above systolic pressure for 5 min. The cuff will then be deflated to induce reactive hyperaemia, whereas PAT recording will be continued. Ten minutes later, the patients will be given a single dose of nitroglycerin (NTG) (0.4 mg, sublingual) to assess endothelium-independent PAT response.

The reactive hyperaemia-PAT data will be analyzed by a computer in an operator-independent manner. As a measure of the extent of reactive hyperaemia, the reactive hyperaemia-PAT index will be calculated as the ratio of the average amplitude of the PAT signal over a 1-min time interval starting 1 min after cuff deflation divided by the average amplitude of the PAT signal of a 3.5-min time period before cuff inflation (baseline); reactive -PAT index values from the study arm will then normalized to the control arm to compensate for potential systemic changes. Hyperaemic response to NTG will be assessed in a similar manner. At first, average PAT signal amplitude of four consecutive 1-min periods starting at 5 min after administration of sublingual NTG (5- to 6-min, 6- to 7-min, 7- to 8-min, and 8- to 9-min interval) will be calculated; PAT response to NTG will then be calculated as the ratio of the PAT amplitude of the 1-min interval during which peak average PAT signal was recorded divided by the amplitude of the PAT signal at baseline (NTG-PAT index).

(v). Cardiopulmonary exercise testing will be determined by means of incremental cycle ergometry. Expired gas analysis will be performed continuously throughout the test with the Innocor System (Innocor, Denmark), which allows determination of VO2 and cardiac output.

Patients will perform a graded maximal bicycle exercise test. After 3 minutes of rest, exercise will begin at a workload of 0 Watts and increase every 3 minutes by 25 Watts until symptom limited maximum. Expired gas analysis will be performed continuously throughout the test with the Innocor System (Innocor, Innovision A/S, Odense, Denmark) which allows determination of VO2 and cardiac output. Peak oxygen uptake will be defined as the highest value of oxygen uptake achieved in the final 20 seconds of exercise. In addition to oxygen uptake [V02], carbon dioxide production [VC0 2], respiratory rate [RR], peak rate pressure product [RPP] and total expiratory volume [VE] will be determined. Anaerobic threshold will be determined from the nadir of the ventilatory equivalent for VO2. Cardiac output will be determined by the inert gas rebreathing method (R), using N2o (blood soluble gas) and SF6 (blood insoluble gas), with concentrations, enriched with o2, of 0.5% and 0.1%, respectively. Tidal volume will progressively increase in the closed circuit to match the physiologic increase. Use of SF6 allows us to measure the volume of lungs, valve and rebreathing bag. N2o concentration decreases during the rebreathing maneuver. Three to four respiratory cycles will be needed to obtain N2o washout.

(vi). Neurohormones: Blood will be drawn for plasma noradrenaline, serum leptin, and adiponectin and plasma cytokines. (a) The quantitative measurement of leptin25-28 in serum performed by using a leptin enzyme immunoassay or ELISA kit29 (DRG Diagnostics, Marburg, Germany), according to the manufacturer's instructions: Briefly, 100µl of diluted leptin conjugate will dispensed into each well of the microtiter plate and incubate at room temperature for 1 h. The contents of the wells will shake out and the wells rinse three times with diluted wash solution. Into each appropriate well were dispensed 50µl of samples (diluted 1:5) and standards at concentrations of 0, 0.8, 1.6, 3.1, 6.2, 12.5, and 25 ng/ml. Fifty microliters of leptin antibody were then dispensed into the center of each well to achieve complete mixing, and the plate will incubate overnight at 4Â°C in a humidity chamber. The contents of the wells will shake out, the wells rinse thrice, and residual droplets will be removed. One hundred microliters of diluted second antibody will dispense into each well and incubate at room temperature for 1.5 h. The contents of the wells will shake out and the wells will be washed three times. One hundred microliters of horseradish peroxidase enzyme complex will dispense into each well and incubate at room temperature for 45 min. Removal and washing of the wells will be repeated before 100µl of tetramethylbenzidine substrate solution will be added and then incubated at room temperature for 20 min. The enzymatic reaction will be terminated by adding 50µl of sulfuric acid stop solution into the center of each well, and the absorbance at 450 nm will determined using an ELISA microtiter plate reader (Tecan, Salzburg, Austria). A standard curve will construct by plotting a graph of the absorbance of each reference standard against its corresponding concentration in nanograms per milliliter. Using the corresponding absorbance to extrapolate the value from the standard curve and multiplying this by the dilution factor of 5 will determine the leptin concentration of each serum sample. (b) Adponetin30-33 levels will be measured by radioimmunoassay by Professor Jill Belch's laboratory. (c) Plasma noradrenaline Blood samples from patients were centrifuged at 4Â°C for 20 minutes, and the separated plasma will immediately frozen and stored at -80Â°C until tested. Plasma noradrenaline (NA) will be measured by high performance liquid chromatography using an electrochemical detector. It is a simplified, sensitive, and reliable method for the determination of NA in plasma.(d) Cytokines: Tumor Necrosis Factor a (TNF- a) ELISA kit will be used for measurement of TNF-a in serum by radioiimunoassay 34-36.

(vii). Physical activity questionnaire; in this study will use Kansas City Cardiomyopathy Questionnaire (KCCQ).

(viii).Endothelial Cell and Blood Collection With use of a 0.021-inch-diameter, J-shaped wire (Daig) inserted through an 18-gauge Angiocath (Becton Dickinson), endothelial cells will be collected from a superficial forearm vein. The wire will transferred to dissociation buffer (0.5% bovine serum albumin, 2 mmol/L EDTA, and 100 _g/mL heparin in phosphatebuffered saline) at 4°C. Cells will be rinsed, fixed in 3.7% formaldehyde, transferred to slides, air dried, and stored at _80°C. Plasma and serum will be separated by centrifugation and stored at _80°C.

ELIGIBILITY:
Inclusion Criteria:

* One hundred patients with Left ventricular Ejection Friction (LVEF) <35% in NYHA class I II III or IV; aged 30-90, attending the CHF clinic will be studied
* Diagnosis of CHF will be based on medical history of exertional dyspneoa, muscle fatigue and/or fluid retention and diminished LVEF (LVEF<35%)
* The diagnosis of ischemic heart disease will be based on documentation of previous myocardial infarction, coronary artery bypass surgery or pathologic findings on coronary angiography. Idiopathic dilated cardiomyopathy will be diagnosed in the absence of a specific etiology for left ventricular dysfunction and on the basis of normal coronary arteries
* All patients should be stable with their treatment and no change in their treatment regimen for > 6 weeks before the study
* Patients with CHF due to coronary artery disease are more likely to have abnormalities in glucose metabolism than are patients with CHF due to idiopathic dilated cardiomyopathy. Therefore, we also plan to study a control group [n=50] of age and sex and BMI matched patients divided into 2 groups 25 with coronary artery disease without heart failure and 25 healthy control. These patients will be identified from the Cardiology Clinics

Exclusion Criteria:

* Patients with decompensated CHF with signs of congestion
* Since the objective of the study is to assess prevalence of insulin resistance in CHF and not CHF secondary to other diseases like diabetes mellitus (DM), patients suffering from DM will be excluded
* Individual found during study cognitively impaired rendering them incapable to take part

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CHF patients were identified from inpatients as well as patients attending outpatient clinics and from the general practice in the community. Diagnosis of CHF was based on the European Society of Cardiology guidelines for CHF (i.e., symptoms of CHF and objective evidence of LV systolic dysfunction). All patients with stable CHF were included in the study. Inpatients with CHF who were hospitalized were also included, except patients with acutely decompensated CHF requiring intravenous therapy. CHF patients with a previous diagnosis of diabetes mellitus were excluded from the study
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2006-08; Primary Completion 2008-07-31 (Actual); Study Completion 2008-07-31 (Actual)

PRIMARY OUTCOMES:
Fasting Insulin Resistance Index | Till end of study
  Fasting insulin resistance index was assessed in a cohort of 129 consecutive CHF patients testing and peripheral endothelial function testing by reactive hyperemia peripheral arterial tonometry (RH-PAT).

CONTACTS AND LOCATIONS:
Overall Officials: Chim C Lang, MD, FRCP, Principal Investigator — University of Dundee, Scotland, UK
Locations (1):
- University of Dundee, Dundee, United Kingdom

REFERENCES:
- [Derived] AlZadjali MA, Godfrey V, Khan F, Choy A, Doney AS, Wong AK, Petrie JR, Struthers AD, Lang CC. Insulin resistance is highly prevalent and is associated with reduced exercise tolerance in nondiabetic patients with heart failure. J Am Coll Cardiol. 2009 Mar 3;53(9):747-53. doi: 10.1016/j.jacc.2008.08.081. PMID 19245964